CLINICAL TRIAL: NCT00987792
Title: CAPRIVI: Community Acquired Pneumonia: Treatment With Avelox® in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14522; AX0801 (Other: Company internal)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Pneumonia
Keywords: Community Acquired Pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Hospitalized patients receiving Avelox according to local drug information

SUMMARY:
The aim of this study is to obtain data from hospitalized Community Acquired Pneumonia (CAP) patients on the disease including disease severity, clinical signs and symptoms and measures used for diagnosis in daily routine practice as well as data on Avelox® including information on the use, effectiveness, treatment outcome, safety and tolerability.

As this is a non-interventional observational study, routine clinical practice is observed. The application of medications follows the normal routines and is decided by the treating physician under recognition of the package insert.

ELIGIBILITY:
Inclusion Criteria:

* Adult hospitalized patients with a diagnosis of CAP (based on local medical practice) and decision taken by the investigator to treat with moxifloxacin and to start treatment with intravenous administration. The local moxifloxacin product information must be considered.

Exclusion Criteria:

* Contraindications stated in the local moxifloxacin product information; warnings and precautions must be considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male hospitalized adult patients scheduled to be treated with moxifloxacin for their CAP and starting treatment with intravenous administration will be documented after the attending physician made the therapeutic decision at his/her discretion.
Sampling Method: Non-Probability Sample
Enrollment: 2595 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the distribution of the CRB-65 severity index at baseline in hospitalized patients suffering from CAP and to whom moxifloxacin (starting with intravenous administration) was prescribed, in countries from South Eastern | At baseline only

SECONDARY OUTCOMES:
Assessment of use of different diagnostic measures in daily routine practice, especially chest radiography and microbiology | 7-14 days
Determination of the proportion of patients treated with moxifloxacin as antibiotic second-line therapy | 7-14 days
Assessment of clinical signs and symptoms before and after therapy with moxifloxacin | 7-14 days
Measurement of moxifloxacin treatment success in terms of effectiveness and outcome | 7-14 days
Evaluation of safety and tolerability of moxifloxacin in hospitalized CAP patients | 7-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Croatia
- Many Locations, France
- Many Locations, Hungary
- Many Locations, Jordan
- Many Locations, Kazakhstan
- Many Locations, Lebanon
- Many Locations, Moldova
- Many Locations, North Macedonia
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Ukraine

REFERENCES:
- [Result] Kuzman I, Bezlepko A, Kondova Topuzovska I, Rokusz L, Iudina L, Marschall HP, Petri T. Efficacy and safety of moxifloxacin in community acquired pneumonia: a prospective, multicenter, observational study (CAPRIVI). BMC Pulm Med. 2014 Jun 30;14:105. doi: 10.1186/1471-2466-14-105. PMID 24975809